CLINICAL TRIAL: NCT02346383
Title: Optimal Stimulation Programming for Spinal Peripheral Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolinas Center for Advanced Management of Pain (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Eugene Mironer, M.D., PI, Carolinas Center for Advanced Management of Pain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7175
Record Dates: First submitted 2013-10-15; First posted 2015-01-27 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain
Keywords: back pain; neuromodulation; spinal peripheral neuromodulation; spinal cord stimulation; postlaminectomy pain syndrome
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Injections, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- program 1 (Active Comparator): preset program - epidural and peripheral lead to cover pain Randomized selection of epidural and/or peripheral lead programs from 3 possible programs
  Interventions: Device: preset program
- program 2 (Active Comparator): preset program - epidural and peripheral lead to cover pain Randomized selection of epidural and/or peripheral lead programs from 3 possible programs
  Interventions: Device: preset program
- program 3 (Active Comparator): preset program - epidural and peripheral lead to cover pain Randomized selection of epidural and/or peripheral lead programs from 3 possible programs
  Interventions: Device: preset program

INTERVENTIONS:
Device: preset program — Change to different present program using epidural and peripheral lead to cover pain
  Other Names: epidural and peripheral lead to cover pain (Spinal Cord Stimulator)

SUMMARY:
To determine the best parameters with various leads to cover back and leg pain and provide best pain relief

DETAILED DESCRIPTION:
Prospective double-blinded trial of patients already implanted with SCS to determine which programming model best controls their back and or leg pain. Baseline visit is 2 weeks after implant. Baseline study data is collected, program #1 is started. The visit @ week 4 collects NRS, changes to program #2. The visit @ week 6 collect NRS, and starts program #3. The visit @ week 8 collects NRS. Subject chooses their preferred program from the previous 3 and uses that for the next 12 weeks. The visit @ week 20 collects NRS.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord stimulator implant within last 3 weeks
* NRS > 6
* at least 22 years old
* patients who agree not to add or increase their pain medications during the study

Exclusion Criteria:

* patients with prior spinal cord stimulators
* pregnancy
* infusion pump
* history of substance abuse or dependency in last 6 months

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Carolinas Center For Advanced Management of Pain, Spartanburg, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Participants were randomized to 1 of 3 programs. Data were collected every 2 weeks at the completion of each program. Participants chose their preferred program from the previous 3 for the next 12 weeks.
Period: Overall Study
Arm/Group | All Study Participants
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (Pain)
Description: 0 (no pain)- 10 (worst pain imaginable)
Time Frame: Weeks 4, 6 and 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Program 1 | Program 2 | Program 3
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 5.2 (1.6) | 5.2 (2.2) | 5.3 (1.6)

2. Secondary Outcome: Percent Pain Relief- Subject Self-reported Percentage of Relief With Each Program.
Description: percentage of pain relief- self report
Time Frame: weeks 4, 6, and 8
Measure: Mean (Standard Deviation); unit: percentage of pain relief
Arm/Group | Program 1 | Program 2 | Program 3
Number analyzed (Participants) | 40 | 40 | 40
percentage of pain relief | 52 (22) | 46 (27) | 46 (21)

ADVERSE EVENTS:
Arm/Group | Program 1 | Program 2 | Program 3
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No